CLINICAL TRIAL: NCT06341842
Title: Study Phase II "Proof of Concept", National Multi-centered. Randomised 1:1, Evaluate Whether Dapagliflozin Reduces Chemotherapy Induced Cardiotoxicity in Participants With Breast Cancer Treated With (Neo-) Adjuvant Anthracycline-based Chemotherapy +/- Trastuzumab
Brief Title: Potential Protective Role of SGLT-2 Inhibitors for Chemotherapy-induced Cardiotoxicity
Acronym: PROTECT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Laura Scelsi, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2022-003377-28
Record Dates: First submitted 2024-03-19; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer
Keywords: cardiotoxicity; Dapagliflozin; SGLT-2; breast cancer; Anthracycline-based chemotherapy; trastuzumab; Asymptomatic CTRCD; Symptomatic CTRCD; ESC Cardio-Oncology Guidelines
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Investigator initiated Phase II "proof of concept", multicentre, randomized 1:1, open label, parallel-groups study, designed to evaluate if dapagliflozin reduces chemotherapy induced cardiotoxicity in participants with breast cancer treated with (neo-) adjuvant Anthracycline-based chemotherapy +/- trastuzumab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active group - Dapagliflozin 10 mg (Experimental)
  Interventions: Drug: Dapagliflozin 10mg Tab
- Control group - Standard of care (No Intervention)

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab — Dapaglifloziin 10 mg 1 tab daily
  Other Names: forxiga 10mg
  Arms: Active group - Dapagliflozin 10 mg

SUMMARY:
The purpose of this study is to evaluate whether dapagliflozin reduces chemotherapy-induced cardiotoxicity in participants with breast cancer treated with (neo-)adjuvant Anthracycline-based chemotherapy +/- trastuzumab. The study aims to describe the efficacy for dapagliflozin as compared to standard of care. Participants will be recruited in participating centers, where they are planning on starting (neo-) adjuvant ACT-based chemotherapy and/or trastuzumab for stage I-III breast cancer.

DETAILED DESCRIPTION:
Anthracyclines (AC) are among the most widely used chemotherapeutic agents and have been shown to be effective in a wide range of tumors, in particular breast cancer. Their clinical effectiveness, however, may be thwarted by the development of cardiotoxicity that negatively affects patients' outcomes and seriously limits their oncological therapeutic opportunities. A subgroup of breast cancer with overexpressed human epidermal growth factor receptor type 2 (HER2), associated with poor prognosis, is now treated with highly effective targeted therapies such Trastuzumab, Pertuzumab, trastuzumab Emtansine (T-DM1), Trastuzumab Deruxtecan. Based on several large-scale trials of adjuvant therapy in breast cancer, the rate of cardiac dysfunction ranged from 7 to 34%, with HF (NYHA class III or IV) rates between 0 and 4%. In the last twenty years several randomized and observational trials tried to study a prophylactic intervention in order to avoid drug-induced cardiotoxicity and the onset of heart failure. A meta-analysis published in 2019 showed a significant, but small, benefit of neurohormonal therapies in reducing decline in LV systolic function among patients undergoing chemotherapy. SGLT-2 inhibitors are a class of drugs primary developed as oral hypoglycemic medications for diabetic patients. In several trials SGLT-2 inhibitors (also known as gliflozins) have reduced HF hospitalization, CV mortality and all-cause mortality to a different extent, suggesting a pleiotropic effect which goes beyond glycemic control since some RCTs have employed these medications in non-diabetic patients. Currently there is a lack of human evidence in the role of these medications to prevent heart failure induced by chemotherapies. Quagliarello et al performed a preliminary cellular studies on mouse cardiomyocytes (HL-1 cell line) exposed to doxorubicin alone or combined to empaglifozin. In preclinical study, empaglifozin increased left ventricle ejection fraction and fraction shortening compared to doxorubicin groups (p < 0.05), prevented the reduction of radial and longitudinal strain after 10 days of treatment with doxorubicin. These findings provides the proof of concept for translational studies designed to reduce adverse cardiovascular outcomes in non-diabetic cancer patients treated with doxorubicin. Recently, Gongora et al conduct a retrospective study to test the cardiac efficacy and overall safety of SGLT2 inhibitors in patients treated with anthracyclines. The authors conclude that SGLT2 inhibitors were associated with lower rate of cardiac events among patients with cancer and DM who were treated with anthracyclines. Additionally, SGLT2 inhibitors appeared to be safe. These data support the conducting of a randomized clinical trial testing SGLT2 inhibitors in patients at high cardiac risk treated with anthracycline.

The PROTECT trial seeks primarily to assess whether the administration of dapagliflozin is associated with a lower rate of asymptomatic and symptomatic CTRCD during 18 months . The key secondary is to assess whether the administration of dapagliflozin is associated with a lower rate of asymptomatic CTRCD during 18 months. Patients will be recruited in participating centers, where they are planning on starting (neo-) adjuvant ACT-based chemotherapy and/or trastuzumab for stage I-III breast cancer. The enrollment will be ongoing for 1 year until the needed number of patients are recruited.

After screening for inclusion and exclusion criteria, patients will be randomized using a web-based system stratified by the use of trastuzumab to: Active group: chemotherapy regimen plus standard of care plus dapagliflozin (10 mg/die) during 18 months; Control group: chemotherapy regimen plus standard of care during 18 months.During follow-up period, if a patient develops asymptomatic or symptomatic systolic disfunction should be treated according to good clinical practice in both arms.

The sample size is computed based on the primary endpoint and makes use of the data reported in the literature. At 18 months, we expect a cumulative incidence of CTRCD of 35% in the control arm, corresponding to an event-free survival rate of 65%. With 316 patients (158 per arm) we will be able to elicit an increase in event-free survival in the dapaglifozin arm up to 80% (hazard ratio, HR 0.52, 78 events) with a power of 80 and type I error (2-tailed) of 5%. This sample size accounts for a 10% dropout rate and is based on the logrank test to compare event-free survivals. For calculation we used the Stata command: power logrank .65 .80, wdprob(.1) power(.80) alpha(0.05)

ELIGIBILITY:
Inclusion Criteria:

* Chemotherapy-naive patients, scheduled for antracycline +/- trastuzumab treatment in the (neo-)adjuvant setting for stage I-III breast cancer.
* Adult women between 18 and 70 years of age
* eGFR>25 ml/min/1.7 mq
* ECOG score 0-2Consent form signed. Female patients of childbearing potential (not surgically sterilized and between menarche and 1 year post menopause) must have a negative result from a serum pregnancy test performed within 7 days of randomization and on the day of first study treatment prior to the initiation of study treatment. Women of childbearing potential must agree to use highly effective contraceptive measures from the time of informed consent through 7 months after last dose of study drug. Women of childbearing potential willing to use highly effective contraceptive measures from the time of informed consent through 7 months after last dose of study drug .

Exclusion Criteria:

* Left ventricular ejection fraction (LVEF) <53%*
* Valvular heart disease.
* Previous malignancy requiring treatment with anthracyclines or chest radiotherapy.
* A life expectancy of ≤12 weeks.
* Currently pregnant (confirmed with positive pregnancy test performed from -7 to -1 days prior to start study drug) or unwilling to adopt highly effective contraceptive method.
* Currently breast-feeding women
* History of hypersensitivity to dapagliflozin or any of the excipients of the product.
* History of Diabetic Ketoacidosis (DKA) requiring medical intervention (e.g. emergency room visit and/or hospitalization) within 1 month prior to enrolment visit.
* Type 1 diabetes mellitus

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2025-04-19 (Estimated); Study Completion 2025-04-19 (Estimated)

PRIMARY OUTCOMES:
Assess whether the administration of dapagliflozin is associated with a lower rate of asymptomatic and symptomatic CTRCD during 18 months during a 18 months follow-up. | baseline, 3 months, 6 months, 12 months and 18 months.
  Change of Left Ventricular Ejection Fraction Global Longitudinal Strain at 3-6-12 and 18 months compared with baseline will be measured using transthoracic echocardiography.

SECONDARY OUTCOMES:
Difference in severe, moderate and mild asymptomatic CTRCD between the two groups during 18 months according to the background therapy with AC with or without TZ and with or without the use of any of ACEi, angiotensin receptor blockers, or b-blockers | baseline, 3 months, 6 months, 12 months and 18 months.
  Change of Left Ventricular Ejection Fraction Global Longitudinal Strain at 3-6-12 and 18 months compared with baseline will be measured using transthoracic echocardiography.
Difference in symptomatic CTRCD between the two groups during 18 months according to the background therapy with AC with or without TZ (subgroup analysis) | baseline, 3 months, 6 months, 12 months and 18 months.
  Change in Left Ventricular Ejection Fraction Global Longitudinal Strain at 3-6-12 and 18 months compared with baseline will be measured using transthoracic echocardiography.
Change from baseline in end diastolic and systolic left ventricular volumes and in left atrial volume during 18 months | baseline, 3 months, 6 months, 12 months and 18 months.
  transthoracic echocardiography.
Change from baseline of at least of one grade of diastolic disfunction (according to ESC guidelines during 18 months. | baseline, 3 months, 6 months, 12 months and 18 months.
  transthoracic echocardiography.
Change in plasma levels of the bio-humoral marker NT-pro-BNP between baseline and follow-up | baseline, 3 months, 6 months, 12 months and 18 months.
  Change in plasma levels of the bio-humoral marker between baseline and follow-up at three, six, twelve and eighteen months: NT-pro-BNP (pg/mL).
Change in plasma levels of the bio-humoral marker hsTNI between baseline and follow-up | baseline, 3 months, 6 months, 12 months and 18 months.
  Change in plasma levels of the bio-humoral marker between baseline and follow-up at three, six, twelve and eighteen months: hsTNI (ng/mL).
Change in plasma levels of the bio-humoral marker CKD-EPI eGFR between baseline and follow-up | baseline, 3 months, 6 months, 12 months and 18 months.
  Change in plasma levels of the bio-humoral marker between baseline and follow-up at three, six, twelve and eighteen months: CKD-EPI eGFR (mL/min/1.7mq).
Change in plasma levels of the bio-humoral marker hsCRP between baseline and follow-up | baseline, 3 months, 6 months, 12 months and 18 months.
  Change in plasma levels of the bio-humoral marker between baseline and follow-up at three, six, twelve and eighteen months: hsCRP (mg/dL).

OTHER OUTCOMES:
Safety Outcomes: TEAE incidence | baseline, 3 months, 6 months, 12 months and 18 months.
  In order to detect adverse events to dapagliflozin investigators should control any difference in the rate of occurrence of Treatment Emergent Adverse Events (TEAE) between the two groups.
Toxicity: renal failure evaluation. | baseline, 3 months, 6 months, 12 months and 18 months.
  Investigators should control decline in eGFR under 25 ml/min/1.7 mq.
Toxicity: hypoglycaemia evaluation | baseline, 3 months, 6 months, 12 months and 18 months.
  Investigators should control the level of glycemia (mg/dL) documenting clinical hypoglycaemic events.
Tolerability: genito-urinary tract infections | baseline, 3 months, 6 months, 12 months and 18 months.
  Investigators should control genito-urinary tract infections (urinalysis).
Tolerability: symptomatic hypotension | baseline, 3 months, 6 months, 12 months and 18 months.
  Investigators should control symptomatic hypotension.
Quality of Life questionaire: EQ-5D-5L | baseline, 18 months.
  Investigators should control quality of life of the patient with a QOL questionaire (EQ-5D-5L).

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Greco A, Quagliariello V, Rizzo G, Tedeschi A, Schirinzi S, Turco A, Galiazzo M, Acquaro M, De Amicis M, Klersy C, Ghio S, Perrone L, Paccone A, Uccello G, Canale ML, Oliva S, Guerra F, De Luca L, Maurea N, Scelsi L. SGLT2i Dapagliflozin in primary prevention of chemotherapy induced cardiotoxicity in breast cancer patients treated with neo-adjuvant anthracycline-based chemotherapy +/- trastuzumab: rationale and design of the multicenter PROTECT trial. Cardiooncology. 2025 Sep 1;11(1):79. doi: 10.1186/s40959-025-00368-9. PMID 40890873